CLINICAL TRIAL: NCT01285089
Title: Prospective French Study on ACQUIred Haemophilia Treatment With Recombinant Factor VIIa (NovoSeven®) A Prospective Observational Study on the Use of NovoSeven® (Activated Recombinant Human Factor VIIa) for the Haemostatic Treatment of Bleeding Episodes in Patients With Acquired Haemophilia
Brief Title: Observational Study on the Use of NovoSeven® for Haemostatic Treatment of Bleeding Episodes in Patients With Acquired Haemophilia
Acronym: ACQUI-7
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: F7HAEM-3856; U1111-1114-8926 (Other: WHO)
Record Dates: First submitted 2011-01-26; First posted 2011-01-27 (Estimated); Last update posted 2014-01-30 (Estimated); Status verified 2014-01

CONDITIONS: Acquired Bleeding Disorder; Acquired Haemophilia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Drug: activated recombinant human factor VII

INTERVENTIONS:
Drug: activated recombinant human factor VII — Data collection of the use of activated recombinant human factor VII observed through real-world treatment practices

SUMMARY:
This study is conducted in Europe. The aim of this prospective, observational study are to describe the different clinical practice and detailed haemostatic management of activated recombinant human factor VII (NovoSeven®) in patients with acquired haemophilia in France. The secondary aim is to assess the primary haemostasis disorder associated with the coagulation disorders, if available.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with acquired haemophilia
* Treated with activated recombinant human factor VII as first line treatment
* Treated with activated recombinant human factor VII after January 2011

Exclusion Criteria:

* Patients with first diagnosis before january 2010 and having a relapse after january 2011
* Known hypersensitivity to NovoSeven®, or to mouse, hamster or bovine protein

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patient diagnosed with acquired haemophilia and treated with at least one injection of activated recombinant human factor VII can be included in the study. The treatment will be performed according the local practice.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2010-12; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Identification of decision criteria to treat patient with activated recombinant human factor VII | Year 3

SECONDARY OUTCOMES:
Number of patients with a control of bleeding | Year 3

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Paris La Défense Cedex, France

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com